CLINICAL TRIAL: NCT06665633
Title: Treatment of U.S. Veterans With Mild Traumatic Brain Injury With Hyperbaric Oxygen Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Alison Bested, Alison C. Bested MD, FRCPC. Associate Professor, Chair Hyperbaric Medicine, Nova Southeastern University, Nova Southeastern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB#: 2021-406
Record Dates: First submitted 2024-07-12; First posted 2024-10-30 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Mild Traumatic Brain Injury; Hyperbaric Oxygen Therapy; Depression
Keywords: Mild Traumatic Brain Injury; Hyperbaric Oxygen Therapy; Brain SPECT Scan; Brodmann Areas; Suicide; Depression
MeSH Terms: conditions — Brain Concussion; Depression; Suicide | interventions — Oxygen; Gases; Inhalation

STUDY DESIGN:
Intervention Model Description: Pilot study - to study the effect of 40 treatments of hyperbaric oxygen therapy using 100% oxygen and increased atmospheric pressure of 1.5 atmospheres for 60 minutes on chronic mild traumatic brain injury with a wait time of at least 6 months or more after the traumatic brain injury occurred in the U.S. Veterans.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment of U.S. Veterans with mild traumatic brain injury with hyperbaric oxygen therapy (Other): Pilot Study - A total of 40 HBOT treatments at 1.5 atmospheres absolute (ATA) for a dive time of 60 minutes, twice a day Monday through Friday. The treatments were separated by an air break of 4 hours on the same day. Measurements of the effectiveness of HBOT in mTBI done before and after HBOT.
  Interventions: Drug: Oxygen 100 % Gas for Inhalation; Device: Hyperbaric Oxygen Therapy Chamber

INTERVENTIONS:
Drug: Oxygen 100 % Gas for Inhalation — Oxygen 100% Gas for Inhalation in Hyperbaric Oxygen Therapy Chamber at 1.5 ATA
  Other Names: Oxygen
Device: Hyperbaric Oxygen Therapy Chamber — Hyperbaric Oxygen Therapy, 40 treatments, at 1.5 ATA and 100% Oxygen

SUMMARY:
Mild traumatic brain (mTBI) injury affects 400,000 U.S. Veterans resulting in physical, cognitive and mental health symptoms. The Department of Defense (DoD) reported 26 suicides a day from mTBI despite ongoing care for the Veterans. The purpose of this pilot research study is to evaluate the effect of treating Veterans suffering from mTBI or persistent post-concussion syndrome with hyperbaric oxygen therapy (HBOT).

DETAILED DESCRIPTION:
In 40 male U.S. Veterans, who have had chronic mTBI for at least six months, the effect of HBOT will be measured in this pilot study with online questionnaires before and after HBOT to measure mental health issues (e.g. depression) and brain function (e.g. memory). The questionnaires will be repeated at 6 and 12 months after HBOT. Brain SPECT (single-photon emission computerized tomography) scans, will measure blood flow to the brain's injured areas before and after HBOT. Quantitative Electroencephalography (QEEG)) will measure brain electrical signals before and after HBOT. An overnight sleep study will measure the quality and stages of sleep pre- and post-HBOT. Blood tests will measure inflammation and cellular mitochondrial function (energy production by the cell) before and after HBOT.

ELIGIBILITY:
Inclusion Criteria:

* A male U.S. Veteran, suffer from mild traumatic brain injury characterized by:

  1. a confused or disoriented state which lasts less than 24 hours
  2. loss of consciousness for up to 30 minutes
  3. memory loss lasting less than 24 hours. In good health prior to mild traumatic brain injury.

Exclusion Criteria:

An individual is ineligible to participate if does not meet the criteria for mild traumatic brain injury and if any of the following apply:

1. Female gender due to small pilot study and hormonal changes in women.
2. Current treated or untreated major depression with psychotic or melancholic features, schizophrenia, bipolar disorder, delusional disorders, dementias of any type, and alcoholism or drug abuse
3. Current heavy use of alcohol or tobacco use (self-report in last 6 months)
4. Current organ failure (as determined by self-report)
5. Current treated or untreated rheumatologic and inflammatory disorders, as determined by medical diagnosis of one or more of the following: osteoarthritis, rheumatoid arthritis, lupus erythematosus, spondyloarthropathies - ankylosing spondylitis and psoriatic arthritis, Sjogren's syndrome, gout, scleroderma, infectious arthritis, and polymyalgia rheumatica
6. Chronic active infections such as HIV, hepatitis B, and hepatitis C (self-report)
7. History of organ transplant (self-report)
8. Current primary sleep disorders such as insomnia, sleep related breathing disorders, etc.

   (self-report)
9. Any allergic disease (self-report) such as allergic asthma
10. Use of medications that could affect immune function (e.g., steroids, immunosuppressants) (self-report)
11. Renal insufficiency
12. Hepatic insufficiency
13. Currently have no exclusionary diagnoses that could reasonably explain the symptoms of their fatiguing illness and their severity, using the exclusion criteria best described in case definition paper for Chronic Fatigue Syndrome (CFS), as described in detail in Reeves, et all 2003, which clarifies exclusionary conditions.
14. History of moderate to severe traumatic brain injury or TBI requiring hospitalization in the past five years.
15. Unstable PTSD or PTSD requiring hospitalization in the past 5 years (stable PTSD is allowed) - this is to reduce the risk of a claustrophobic triggering of PTSD symptoms.

    (limits generalizability of results to mild/moderate stable PTSD)
16. Are scheduled for surgery during time of hyperbaric oxygen treatments.

Contraindication for HBOT Therapy: untreated collapsed lung.

Relative contraindications for HBOT Therapy: Includes pulmonary diseases including chronic obstructive lung disease, an air blister in the lung that appears on a chest radiograph but does not result in symptoms, upper respiratory or sinus infections, recent ear or thoracic surgery, uncontrolled fever, and claustrophobia. However, these are relative contraindications, which should not deter clinicians from using HBOT to treat patients with severe neurological injuries or other life or limb threatening conditions. The adverse effects of several medications are thought to be increased by HBOT, including bleomycin and doxorubicin. Other exclusions from participation includes pregnancy and participating in another interventional clinical trial of an investigational therapy within 30 days of consent or scheduled for surgery.

Contraindication for brain SPECT scan: Known allergy to radioactive tracer material.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Brain SPECT Scan | pre- HBOT and 4 weeks after HBOT
  A brain SPECT scan is a type of imaging test that uses a radioactive substance and a special camera to create 3D pictures of the brain. It shows which areas of the brain are functioning the best or worst and how well the blood flows in the brain. The blood flow to the brain was measured pre- and post-HBOT. An infusion of a radioactive tracer, 30 millicurie (mCi) of Tc99m-Ceretec, was injected into the Veteran's IV site. The veteran was placed under the gamma scintillation camera (Siemens E-cam Dual Head) with a low-energy, high-resolution collimator and SPECT images were recorded using the NeuroGam Software Analysis for the numerical calculation of the mean blood flow value for each of the Brodmann Areas - which are the functional areas in the brain.

SECONDARY OUTCOMES:
Beck Anxiety Inventory | pre- HBOT and 1, 6. 12 months after HBOT
  The Beck Anxiety Inventory (BAI) is a validated 21-item self-report questionnaire used to assess the severity of anxiety symptoms. Higher scores indicate more severe symptoms. A score of 0-7 indicates minimal anxiety, 8-15 mild anxiety, 16-25 moderate anxiety, and 26-63 severe anxiety.
Beck Depression Inventory II | pre- HBOT and 1, 6. 12 months after HBOT
  The Beck Depression Inventory is a validated self-report questionnaire that indicates the severity of depressive symptoms. Scores are typically categorized as minimal (0-13), mild (14-19), moderate (20-28), or severe (29-63) depression, with higher scores indicating more pronounced symptoms.
Brief Pain Inventory | pre- HBOT and 1, 6. 12 months after HBOT
  It is a validated self-report questionnaire used to assess pain in patients. It measures the intensity of pain (severity) and how it interferes with daily activities (interference). It is scored by calculating the mean of the items for pain severity and pain interference, each on a scale of 0-10. The higher the score, the more intense the pain and the more it interferes with daily activities.
Traumatic Brain Injury Screening Tool | pre- HBOT
  Criteria for Mild Traumatic Brain Injury:
  * Confused/disoriented state that lasts less than 24 hours
  * Loss of consciousness for up to 30 minutes
  * Memory loss lasting less than 24 hours
  * Excluded severe TBI with skull penetrating injury, brain hemorrhage Other cognitive difficulties include feeling dazed, groping for words, and having problems with attention, concentration, processing speed, planning, reasoning, and abstract thinking. Physical symptoms include headache, nausea, vomiting, drowsiness, fatigue, dizziness, loss of balance, blurred vision, unrefreshed sleep, sensitivity to light or sound, tinnitus, and alteration of taste or smell. Some patients also experience mental health symptoms including anxiety, depression, post-traumatic stress disorder, and suicide ideation
Davidson Trauma Scale | pre- HBOT and 1, 6. 12 months after HBOT
  It is a validated 17-item self-report questionnaire used to assess the severity of post-traumatic stress disorder (PTSD) symptoms. The total score, which can range from 0 to 136. Higher scores indicate more severe PTSD symptoms.
Functional Capacity Scale | pre- HBOT and 1, 6. 12 months after HBOT
  Self-report scale from 0 to 10 to measure the severity of fatigue and cognitive ability. Better energy and cognitive function is reflected in a higher number.
Pittsburgh Sleep Quality Index | pre- HBOT and 1, 6. 12 months after HBOT
  It is a validated self-report questionnaire that assesses sleep quality over a one-month time interval. The sum of these component scores yields a global PSQI score, ranging from 0 to 21, with higher scores indicating poorer sleep quality. A global PSQI score greater than 5 is generally considered indicative of poor sleep quality.
The Quick Environmental Exposure and Sensitivity Inventory (QEESI) | pre- HBOT and 1, 6. 12 months after HBOT
  It is a validated self-report questionnaire that helps researchers, doctors, and their patients identify individuals with multiple chemical intolerances and their responses to the chemicals. The score is 0-10 with the higher score indicating a worse response to chemical exposures.
Short-Form 36 Health Survey | pre- HBOT and 1, 6. 12 months after HBOT
  It is a validated questionnaire used to measure health-related quality of life. It has eight scaled scores, each ranging from 0 to 100, with lower scores indicating more disability and higher scores indicating less disability. The eight scales are physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health.
Quantitative Electroencephalography | pre- HBOT and 1 month after HBOT
  It measures the electrical activity in the form of brain wave patterns of the brain. It is called brain mapping and measures quantitative metrics related to cognitive brain functions. It quantitatively measures the delta, theta, alpha and beta bands.
Overnight Sleep Study | pre- HBOT and 1 month after HBOT
  The Cerebra software system is used at home and measures the sleep for one night and includes measuring the percentage of oxygen saturation in the blood as % oxygen using a pulse oximeter, measures heart rate in beats per minute on ECG, breathing rate - measures breathes per minute, limb movement - records leg movement per hour, measures total minutes of time spent snoring, measures the sleep position - in minutes of time spent on back or sides, and measures amount of minutes on EEG brain waves in the different sleep stages including: non-rapid eye movement (NREM) sleep, rapid eye movement (REM) sleep, and stages III/IV sleep. A final report summarizes the sleep study findings.
Measure Blood Markers of Inflammation | pre- HBOT and 1 month after HBOT
  Measure 18 blood cytokines using Q-Plex Array. Measures levels of Tumor Necrosis Factor-1, Interleukin-1a,Interleukin-1b, Interleukin-2, Interleukin-4, Interleukin-5, Interleukin-6,Interleukin -8, Interferon gamma, Interleukin12p70, Interleukin-13, Interleukin-23, Interleukin-15, Interleukin-17, Interleukin-10, Tumor Necrosis Factor alpha, Tumor Necrosis Factor-Receptor II, Tumor Necrosis Factor beta. All cytokines were measured in picograms/milliliter and measured in the Multiplex Cytokine Analyzer. All of the individual cytokines were compared to normal, high, and low controls.
PTSD Checklist - Stressor Specific Version (PCL-S) | pre- HBOT and 1 month after HBOT
  The PCL is a validated 17-item self-report measure of the DSM-IV symptoms of PTSD. Respondents rate how much they were "bothered by a symptom" on a 5-point scale ranging from 1 ("not at all") to 5 ("extremely"). A higher score indicates the more severe outcome. A score between 31 and 33 is often used as a cut-off score to indicate probable PTSD with 80 the maximum score.
Clinical Criteria for Traumatic Brain Injury Severity | pre- HBOT and 1 month after HBOT
  Clinical Criteria: Mild, Moderate, Severe.
  Structural Imaging: Normal, Normal or abnormal, Normal or Abnormal.
  Loss of Consciousness: < 30 minutes, 30 minutes to 24 hours, > 24 hours.
  Alteration of Consciousness/Mental State: A moment to 24 hrs. > 24 hours > 24 hours.
  Post-traumatic Amnesia: 0-1 day, > 1 and < 7 days, > 7 days.
Mitochondrial Function | pre- HBOT and 1 month after HBOT
  Mitochondrial function is measured in the peripheral blood mononuclear cells (PBMCs) using the Seahorse™ Assay. The PBMCs reflect functioning of the brain's neurons and will assess if there is mitochondrial repair after hyperbaric oxygen therapy.
Measure DNA Repair | pre- HBOT and 1 month after HBOT
  DNA repair measured by measuring Nucleotide Excision Repair in peripheral blood mononuclear cells (PBMCs), which is a reflection of what is occurring in the brain's neurons and will assess if there is DNA repair after hyperbaric oxygen therapy. .
Neurocognitive Index | pre- HBOT and 1, 6. 12 months after HBOT
  It is the average of five domain scores: Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention , and Cognitive Flexibility ; representing a form of a global score of neurocognition. Scores range from less than 70, very low, to greater than 109, above average.
Composite Memory | pre- HBOT and 1, 6. 12 months after HBOT
  Questionnaire measures the ability to recognize, remember, and retrieve words and geometric figures. Scores range from less than 70, very low, to greater than 109, above average.
Verbal Memory | pre- HBOT and 1, 6. 12 months after HBOT
  Questionnaire measures the ability to recognize, remember, and retrieve words. Scores range from less than 70, very low, to greater than 109, above average.
Visual Memory | pre- HBOT and 1, 6. 12 months after HBOT
  Questionnaire measures the recognition memory for abstract figures or shapes. Scores range from less than 70, very low, to greater than 109, above average.
Finger Tapping | pre- HBOT and 1, 6. 12 months after HBOT
  Online computer test process that measures motor speed and fine motor control. Scores range from less than 70, very low, to greater than 109, above average.
Symbol Digit Coding | pre- HBOT and 1, 6. 12 months after HBOT
  Online computer test process that measures complex information, processing accuracy, complex attention, visual-perceptual speed, and information processing speed. Scores range from less than 70, very low, to greater than 109, above average.
Stroop Test | pre- HBOT and 1, 6. 12 months after HBOT
  Online computer test process that measures simple reaction time, complex reaction time, Stroop reaction time, inhibition/disinhibition, and frontal or executive skills. Scores range from less than 70, very low, to greater than 109, above average.
Shifting Attention | pre- HBOT and 1, 6. 12 months after HBOT
  Online computer test process that measures the ability to shift from one instruction set to another quickly and accurately. Scores range from less than 70, very low, to greater than 109, above average.
Continuous Performance | pre- HBOT and 1, 6. 12 months after HBOT
  Online computer test process that measures vigilance or sustained attention or attention over time. Scores range from less than 70, very low, to greater than 109, above average.
Perception of Emotions | pre- HBOT and 1, 6. 12 months after HBOT
  Questionnaire measures how well a subject can perceive and identify specific emotions. Scores range from less than 70, very low, to greater than 109, above average.
Non-Verbal Reasoning | pre- HBOT and 1, 6. 12 months after HBOT
  Questionnaire measures how well a subject can perceive and understand the meaning of visual or abstract information and recognizing relationships between visual-abstract concepts. Scores range from less than 70, very low, to greater than 109, above average.
4-Part Continuous Performance | pre- HBOT and 1, 6. 12 months after HBOT
  It is a four-part online computer test that measures a subject's working memory and sustained attention. Scores range from less than 70, very low, to greater than 109, above average.

CONTACTS AND LOCATIONS:
Overall Officials: Alison C Bested, MD FRCPC, Principal Investigator — Nova Southeastern University
Locations (1):
- Nova Southeastern University, Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
Will need time from data support person to help with data sharing.